CLINICAL TRIAL: NCT04458675
Title: A Prospective, Multicenter, Randomized, Single Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Vibrant Capsule vs. Vibrant Placebo for the Treatment of Chronic Idiopathic Constipation (CIC)
Brief Title: Efficacy and Safety of Vibrant Capsule vs. Vibrant Placebo for the Treatment of Chronic Idiopathic Constipation (CIC)
Acronym: CIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vibrant Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 250CLD
Record Dates: First submitted 2020-06-09; First posted 2020-07-07 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — Equipment and Supplies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active (Experimental): Active capsule
  Interventions: Device: Vibrant capsule
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Device: Vibrant capsule — The capsule vibration mechanically stimulates the inner wall of the GI and stimulates motility
  Other Names: medical device
  Arms: Active
Drug: Placebo — A biodegradable capsule, which visually similar to the Vibrant active capsule
  Other Names: control
  Arms: Placebo

SUMMARY:
The was performed to assess the safety and efficacy of the vibrant capsule vs. placebo for the treatment of subjects with functional Constipation.

DETAILED DESCRIPTION:
Visit 1 -Screening: Subjects will be screened to the study at the screening visit, PAC-QOL questionnaire will be completed and subject will have a run-in time for a period of 2-3 weeks, assuring 14 consecutive days of eDiary with an average of < 3 SBM per week.

Visit 2 - Baseline: After the run-in period, the subjects will return and eligibility will be re-assessed. Subjects will be randomized to either Vibrant or Vibrant placebo for a treatment period of 8 weeks. Subjects, in both arms, will have their first administration of Vibrant capsule / Vibrant placebo on site at the day of baseline visit and will be instructed on their treatment administration at home and will be requested to ingest the capsules at a specific time of the day. At baseline, subjects will also be trained on how to use the base unit at home.

Subjects will be instructed to complete a simple subject eDiary each day throughout the duration of the study (including the run-in period).

The eDiary will include questions on:

* Daily BM, SBM, CSBM
* Change of their diet, if applicable (NOTE: the protocol will not ask/require the subjects to change anything in his/her diet)
* Change in sympotms as: brisol stool consistancy, straining, bloating, and the other questions in the eDiary
* Medication
* AE (including diarhrea)

The first 2 weeks of treatment will be considered as a subjects' training period.

Visit 3 -after 4 weeks of treatment - an on site visit will take place to evaluate subject's safety and treatment efficacy and additional capsule dispencing.

Visit 4 Final visit -after another 4 weeks of treatment - an on site visit will take place to evaluate subject's safety and treatment efficacy and collect the base unites and remaning capsules. PAC-QOL, Ease of use and TSQM questionnaires will be completed.

During the entire study period, data reporting will be done on an electronic Case Report Form (eCRF) and an eDiary.

Subjects will be asked to refrain from taking any medication or supplement to relieve their constipation, during the entire study period.

Subjects will receive phone calls at least once a week and subject compliance will be monitored throughout the 8 weeks of the study.

Subjects will be authorized to use rescue medication after 3 consecutive days without a bowel movement.

Data about time of activation of the capsules will be automatically registered and transmitted by the base unit for Vibrant capsules

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 22 years and older
2. Subjects with Chronic Idiopathic Constipation (CIC) according to Rome III criteria and who have not experienced relief of their symptoms from available therapies (osmotic and stimulant laxatives used for at least one month at recommended dose)
3. Subjects with an average of <3 Spontaneous Bowel Movements (SBM) per week
4. Normal colonoscopy performed within 5 years prior to study participation, unless the subjects are <50 years old and without alarm signs and/or symptoms
5. Subject signed the Informed Consent Form (ICF)
6. Female subjects must have a negative blood pregnancy test during screening, confirmed by a negative urine pregnancy test during baseline and must not be lactating prior to receiving study medication. For females of child-bearing potential, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. All other female subjects must have the reason for their inability to bear children documented in the medical record [i.e., tubal ligation, hysterectomy, or post-menopausal (defined as a minimum of one year since the last menstrual period)]; in these circumstances, a pregnancy test will not be necessary

Exclusion Criteria:

1. History of complicated/obstructive diverticular disease
2. History of intestinal or colonic obstruction, or suspected intestinal obstruction.
3. History of significant gastrointestinal disorder, including any form of inflammatory bowel disease or gastrointestinal malignancy (celiac disease is accepted if the subject has been treated and is in remission)
4. History of gastroparesis
5. Use of any of the following medications:

   * Medications that may affect intestinal motility, prokinetics, anti-Parkinsonian medications, opiates, opioids, calcium-channel blockers, aluminum/magnesium hydroxide
   * With the exception of antidepressants, thyroid or hormonal replacement therapy, when the subject has been on a stable dose for at least 3 months prior to enrollment.
6. Clinical evidence of significant respiratory, cardiovascular, renal, hepatic, biliary, endocrine, psychiatric or neurologic disease.
7. Presence of cardiac pacemaker or gastric electrical stimulator.
8. History of, or current eating disorders, such as anorexia, bulimia, or compulsory overeating.
9. Diagnosis of mega-rectum or colon, congenital anorectal malformation, clinically significant rectocele, history of intestinal resection (with an exception for appendectomy, cholecystectomy and inguinal hernia repair), history of bariatric surgery or evidence of any structural abnormality of the gastrointestinal tract that might affect transit
10. History of Zenker's diverticulum, dysphagia, Barrett's esophagus, esophageal stricture or achalasia
11. Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs): chronic use is defined as taking full dose NSAIDs more than three times a week for at least six months. Subjects on cardiac doses of aspirin may be enrolled in the study
12. Subjects with pelvic floor dysfunction/defecatory disorder, based on subject history
13. Participation in another clinical study within one month prior to screening.
14. Women who are pregnant or lactating
15. Use of any medication for constipation relief during the study, except as rescue medication, as indicated by study rules
16. Inability to use an electronic daily Diary (on a computer, phone application, tablet or other electronic device) to report bowel movements, symptoms and medication usage
17. Subject participated in a previous Vibrant study
18. Any other condition which in the opinion of the investigator may adversely affect the safety of the subject or would limit the subject's ability to complete the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tal Malina, B.SC MBA, Study Director — tal.m@vibrantgastro.com
Locations (1):
- Health Research of Hampton Roads, Newport News, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Placebo
Started | 31 | 28
Completed | 31 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 31 | 28 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.91 (11.87) | 46 (14.95) | 46 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 57
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 15 | 9 | 24
  Hispanic or Latino | 4 | 10 | 14
  Black or African American | 11 | 8 | 19
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 31 | 28 | 59
Duration of constipation [Mean (Standard Deviation); unit: years] | 18.06 (13) | 21.36 (12.32) | 19.62 (12.70)

OUTCOME MEASURES:

1. Primary Outcome: CSBM1 Success Rate
Description: The number of subjects with an increase from the run-in period of at least one weekly Complete Spontaneous Bowel Movement (CSBM) during at least 6 of the 8 weeks of treatment
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 31 | 28
Participants | 9 | 8

2. Primary Outcome: CSBM2 Success Rate:
Description: The number of participants with an increase from the run-in period of at least two weekly Complete Spontaneous Bowel Movements (CSBM) during at least 6 of the 8 weeks of treatment
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 31 | 28
Participants | 7 | 5

ADVERSE EVENTS:
Time Frame: The Safety reporting conducted throughout the treatment period (8 weeks)
Arm/Group | Active | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/28
Other Adverse Events (participants affected / at risk) | 6/31 | 8/28
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=31) | Placebo (N=28)
Diarrhea (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Other (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Permission to use study data is required

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT04458675/Prot_SAP_000.pdf